CLINICAL TRIAL: NCT05901090
Title: Comparing the Effects of Modified Thoracoabdominal Nerve Block Through Perichondrial Approach (M-TAPA) and Transerversus Abdominis Plane Block (TAP) on Postoperative Pain Scores and Total Analgesic Consumption in Patients Ongoing Total Abdominal Hysterectomy
Brief Title: Comparing the Effects of M-TAPA and TAP Block on Postoperative Analgesia in TAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Assisstant Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: M-TAPA vs TAP block on TAH
Record Dates: First submitted 2023-06-01; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Pain
Keywords: m-tapa; tap block; total abdominal hysterectomy; regional anesthesia; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- M-TAPA block (Active Comparator): Patients had bilateral M-TAPA block with 0.25% bupivacaine (total volume of 40 ml) at the end of the surgery for postoperative pain control.
  Interventions: Other: M-TAPA block
- TAP block (Active Comparator): Patients had bilateral TAP block with 0.25% bupivacaine (total volume of 40 ml) at the end of the surgery for postoperative pain control.
  Interventions: Other: TAP block
- Control (No Intervention): Control group patients were not subjected to any block or local infiltration anesthesia. Their postoperative pain was relieved with tramadol (intravenous) administration.

INTERVENTIONS:
Other: M-TAPA block — Following sterile conditions for bilateral M-TAPA block application, the transducer was inserted on the chondrium in the sagittal plane at the 9-10th rib level. Subsequently, a deep angle was created with the probe for visualization of the underside of the costochondrium. The sonovisible needle tip was placed just below the chondrium and saline (5 ml) was injected for site confirmation. After the confirmation, 20 ml of 0.25% bupivacaine was administered for each group for a total of 40 ml of local anesthetic. Blocks were applied using an 80 mm sonovisible needle with a 6-10 MHz linear probe under the guidance of a portable ultrasound. M-TAPA block with the same standard technique and drug dose was applied to the contralateral side for each group of M-TAPA patients.
  Other Names: Modified thoracoabdominal nerve block through perichondrial approach
  Arms: M-TAPA block
Other: TAP block — After the necessary sterilization conditions were established, the linear ultrasound probe was sterilely coated and placed in the middle of the iliac crest with the end limit of the ribs. Starting with skin, the layers in descending order, subcutaneous adipose tissue, external oblique muscle, internal oblique muscle, transversus abdominis muscle, and peritoneum were identified. As the tip of the 80 mm sonovisible needle passed through the muscular layers and fascia, a fascial click was felt and the needle was advanced with ultrasound in a controlled manner. After receiving the second click sensation (passage of the fascia of the internal oblique muscle), the location of the needle was fixed and frequently aspirated and applied to the plane so that 20 ml of 0.25% bupivacaine was applied to each side. (40 ml in total)
  Other Names: Transversus abdominis plane block
  Arms: TAP block

SUMMARY:
Aim is to compare the postoperative analgesic efficacy of M-TAPA block and TAP block and their effect on opioid consumption in patients undergoing open total abdominal hysterectomy (TAH) surgery.

DETAILED DESCRIPTION:
There were three randomized groups: Group M (M-TAPA block) (n=15), Group T (TAP block) (n=15) and Group C (no block) (n=15). All patients had standard general anesthesia. Group M had bilateral M-TAPA block with 0.25% bupivacaine (total volume of 40 ml) at the end of the surgery. Group T patients had TAP block with 0.25% bupivacaine (total volume of 40 ml) at the end of the surgery. Group Control had only tramadol for postoperative pain. Numerical rating scale (NRS) was used to assess postoperative pain on 1st, 6th, 12th and 24th hour after the surgery. Total tramadol consumption was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 35 years of age who underwent open total abdominal hysterectomy under general anesthesia and were American Society of Anesthesiologists (ASA) I-II-III according to the ASA risk classification.

Exclusion Criteria:

* Patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with local anesthetic drug allergies,
* patients undergoing laparoscopic surgery,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Comparing the numerical rating scale scores | Postoperative 24 hours
  Numerical rating scale is used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Comparing total tramadol consumption | Postoperative 24 hours
  Postoperative analgesic need

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Gündoğdu, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)